CLINICAL TRIAL: NCT04917562
Title: Refractive Transepithelial Photo-keratectomy (T-PKR) Without Addition of Mitomycin-C in High Myopia: a Retrospective Study of 69 Eyes
Brief Title: Refractive Transepithelial Photo-keratectomy (T-PKR) in High Myopia
Acronym: TEPEHERKAHM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-03-Obs-CHRMT
Record Dates: First submitted 2021-05-21; First posted 2021-06-08 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2021-05

CONDITIONS: Ophthalmopathy; Myopia; Keratopathy
Keywords: transepithelial photorefractive keratectomy; high myopia; mitomycin-C; corneal haze; efficacy; predictibility
MeSH Terms: conditions — Eye Diseases; Myopia; Corneal Opacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the anatomical and refractive parameters following a single-step transepithelial photo-refractive keratectomy (T-PRK) without the addition of mitomycin-C for the treatment of high myopia of 6 diopters or more.

DETAILED DESCRIPTION:
In this retrospective study, 69 high myopic eyes of 6 diopters or more were treated in 38 patients by Trans-PRK with the SCHWIND Amaris 500E® excimer laser platform without the use of mitomycin-C. Several outcomes are measured in treated patients, such as postoperative uncorrected visual acuity (UCVA), best spectacle corrected visual acuity (BSCVA), efficacy, safety and predictability of the procedure, as well as corneal haze measurement. The patients are followed-up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years,
* myopic sphere of -6 diopters or more,
* astigmatism less than 3 diopters,
* stable myopia not progressing for more than one year

Exclusion Criteria:

* age <18 years,
* myopic sphere less than -6 diopters,
* astigmatism greater than 3 diopters,
* progressive myopia (variation of more than 0.5 diopters over one year),
* abnormal corneal topography or the presence of manifest keratoconus,
* pre-existing eye pathology,
* history of eye surgery,
* active inflammatory or infectious eye disease,
* dermatological disease or systemic connectivitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective study conducted on the eyes of patients with high myopia (less than or equal to -6 diopters) associated or not with astigmatic less than 3 diopters operated by Trans-PRK with the SCHWIND Amaris 500E platform (SCHWIND eye-tech-solutions GmbH, Kleinostheim, Germany) in the CHR Metz-Thionville between January 1, 2018 and January 1, 2020
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative uncorrected visual acuity (UCVA) at week 1 | Week 1
  Postoperative uncorrected visual acuity (UCVA) (logMAR)
Postoperative best spectacle corrected visual acuity (BSCVA) at week 1 | Week 1
  Postoperative best spectacle corrected visual acuity (BSCVA) (logMAR)
Postoperative uncorrected visual acuity (UCVA) at month 1 | Month 1
  Postoperative uncorrected visual acuity (UCVA) (logMAR)
Postoperative uncorrected visual acuity (UCVA) at month 3 | Month 3
  Postoperative uncorrected visual acuity (UCVA) (logMAR)
Postoperative best spectacle corrected visual acuity (BSCVA) at month 1 | Month 1
  Postoperative best spectacle corrected visual acuity (BSCVA) (logMAR)
Postoperative best spectacle corrected visual acuity (BSCVA) at month 3 | Month 3
  Postoperative best spectacle corrected visual acuity (BSCVA) (logMAR)

SECONDARY OUTCOMES:
Visual acuity efficacy index | 3 months
  The efficacy of the procedure was defined by the proportion of eyes with uncorrected visual acuity at 3 months greater than or equal to Log MAR 0.1 (or 8/10 on a decimal scale). The efficacy index was defined as the ratio between the mean uncorrected visual acuity at 3 months and the best corrected visual acuity preoperatively. A threshold of 80% was required to consider the surgery successful.
Visual acuity safety index | 3 months
  The safety of the procedure was defined as the proportion of eyes that lost 2 or more lines of visual acuity compared to the best preoperative corrected visual acuity.
  The safety index was defined as the ratio between the best corrected visual acuity 3 months postoperatively and the best corrected visual acuity preoperatively. An 80% threshold was chosen to consider the procedure safe.
Predictability | 3 months
  Predictability was defined as the percentage of eyes having reached target refraction (± 0.5D) at the end of follow-up (3 months).
Postoperative corneal haze measurement at week 1 | Week1
  Corneal haze assessment was performed at each follow-up visit and reported on the Fantes scale
  * Grade 0: absence of corneal haze.
  * Grade 1: corneal fog that does not prevent the visibility of details of the iris
  * Grade 2: slight fading of details of the iris
  * Grade 3: pronounced erasure of details of the iris and lens
  * Grade 4: complete opacification of the stroma preventing access to the anterior chamber
Postoperative corneal haze measurement at month 1 | Month 1
  Corneal haze assessment was performed at each follow-up visit and reported on the Fantes scale
  * Grade 0: absence of corneal haze.
  * Grade 1: corneal fog that does not prevent the visibility of details of the iris
  * Grade 2: slight fading of details of the iris
  * Grade 3: pronounced erasure of details of the iris and lens
  * Grade 4: complete opacification of the stroma preventing access to the anterior chamber
Postoperative corneal haze measurement at month 3 | Month 3
  Corneal haze assessment was performed at each follow-up visit and reported on the Fantes scale
  * Grade 0: absence of corneal haze.
  * Grade 1: corneal fog that does not prevent the visibility of details of the iris
  * Grade 2: slight fading of details of the iris
  * Grade 3: pronounced erasure of details of the iris and lens
  * Grade 4: complete opacification of the stroma preventing access to the anterior chamber
postoperative spherical equivalent | 3 months
  Percent of postoperative spherical equivalent D (SD)
Postoperative refractive astigmatism at +/- 0.5D of target | 3 months
  Percent of eyes within +/- 0.5D of target
Postoperative refractive astigmatism at +/- 1.0D of target | 3 months
  Percent of eyes within +/- 1.0D of target
Complications | Up to 3 months
  Percent of postoperative infections or epithelial healing
Patient sex | Before surgery
  Sex ratio Men/Women (percent)
Patient age | Before surgery
  Age (years)
Preoperative Myopia | Before surgery
  Myopia (Diopters)
Preoperative Astigmatism | Before surgery
  Astigmatism (Diopters)
Preoperative Spherical equivalence | Before surgery
  Spherical equivalence (Diopters)
Preoperative best spectacle corrected visual acuity | Before surgery
  BSCVA (logMAR)
Preoperative Keratometry | Before surgery
  Keratometry (dipoters)
Preoperative central corneal thickness | Before surgery
  central corneal thickness (µm)
Preoperative optical and transition zones | Before surgery
  Optical and transition zones (mm)
Preoperative total ablation thickness | Before surgery
  Total ablation thickness (µm)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc PERONE, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- Centre Hospitalier Metz Thionville, Metz, France